Evaluation of Pain Quality in Young Swimmers Suffering from Myofascial Pain Syndrome Using Lidocaine Phonophoresis: A Pilot Study in Physical Therapy Rehabilitation Center in Egypt

## **Brief description**

Myofascial pain syndrome (MPS) is characterized by pain and accompanying muscle spasm, referred pain patterns, stiffness, restricted range of motion caused by trigger points on constricted fibers of the skeletal muscles or fasciae. Myofascial pain syndrome is the most common reason of neck and shoulder pain.

The main goal of MPS treatment is to break down the vicious circle of pain spasm and release of trigger points. Various physical therapy modalities such as trigger point injection, stretching-spray technique, heat packs, and transcautaneous electrical nerve stimulation are used for the treatment of MPS.

Therapeutic ultrasound was developed and widely used in the daily practice of physical therapy and sport medicine for the treatment of a variety of acquired and traumatic conditions in overuse injuries. Phonophoresis is believed to accelerate functional recovery by decreasing pain and promoting healing and it has been used to administer various drugs mainly local anesthetics.

Alyhough many different modalities are available to treat MPS especially therapeutic ultrasound and there was lack of research works that investigated the effect of phonophoresis with local anesthetics on myofascial trigger points, so it was of value to compare between the effect of lidocaine phonophoresis and pulsed ultrasound on MPS in treatment of neck pain in youth swimmers using Pain Quality Assessment Scale as a tool of pain quality evaluation.

## Corresponding author

Mohamed Abdel-Moneim Abo-EL-Roos

Email address: mohamed.aboelros@pt,.ninu.edu.eg

| I am father / mother ofresearch program under the direct | | conse | nt to participate in a |
|---|---|---|---|
| A thorough description of the promay withdraw my consent and diswithout prejudice to me. | * | | |
| Date | Participant | | |
| If illiterate | | | |
| A literate witness must sign (i participant and should have no co illiterate should include their thun | onnection to the research t | | - |
| I have witnessed the accurate potential participant, and the questions. I confirm that the inc | e individual has had | the o | opportunity to ask |
| Print name of witness | A | ND | Thumb print of |
| participant Signature of witness Date | | | |
| Day/month/year | | | |

Statement by the researcher/person taking consent.

I have accurately read out the information sheet to the parent of the potential participant, and to the best of my ability made sure that the person understands that the following will be done:

1.

2.

I confirm that the parent was given an opportunity to ask questions about the study, and all the questions asked by him/her have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily.

Print Name of Researcher/person taking the consent\_\_\_\_\_